CLINICAL TRIAL: NCT00465296
Title: Ppar-Gamma EliminAtes Restenosis Longevity Study: PEARLS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding Discontinued
Sponsor: Medstar Health Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PEARLS
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2007-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
The primary objective of this clinical trial is to assess the efficacy of rosiglitazone on bare metal stent (BMS) in-stent restenosis measured as late lumen loss in patients with metabolic syndrome.

The secondary parameter for evaluation of efficacy is binary restenosis.

The tertiary objective will be to assess the effect of rosiglitazone on major cardiac events (MACE; death, MI, CABG, and target vessel revascularization). The occurrence of in-stent restenosis for patients with metabolic syndrome who receive a DES in a non-target lesion will be assessed angiographically at 9 months.

DETAILED DESCRIPTION:
This is a prospective, multicenter, double blind, randomized clinical trial of patients who present to the catheterization laboratory for PCI (elective or setting of ACS) and receive at least one bare metal stent.

Patients will be randomized on a 1:1 basis to receive either rosiglitazone or placebo for 9 months. Patients will be followed for 9 months post procedure. All patients will be required to have a repeat angiogram with optional IVUS analysis at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age >/=18 years;
* Patients must meet MS definition, which means that each patient must meet at least 3 of listed requirements of MS:

  * A waist circumference of 40 inches or more for men and 35 inches or more for women (measured across the belly);
  * A blood pressure of 130/85 mm Hg or higher;
  * A triglyceride level 150 mg/dl or above;
  * A fasting blood glucose level greater than 110 mg/dl , but less than 126; and/or
  * A high density lipoprotein level (HDL) less than 40 mg/dl (men) or under 50 mg/dl (women).
* Patients eligible for PCI;
* Patients must receive at least one bare metal stent;
* The patient has stable or unstable angina with clinical evidence of ischemia (ECG, exercise test, etc.); and/or
* The patient is able and willing to conform to the requirements of the study including repeat angiographic follow-up at 9 months, and voluntarily signs an Informed Consent.

Exclusion Criteria:

* • Patient has experienced an ST-segment elevation myocardial infarction within the preceding 48 hours; Patient must have CPK and CK-MB <3 times upper limit of normal at the time of angioplasty and enrollment;

  * Previously diagnosed with either type 1 or type 2 diabetes and controlling glucose by one or a combination of the following treatments: diet, oral anti-diabetic agents, or insulin;
  * Patient had or plans to have CABG within 9 months;
  * Ejection fraction <35%; class III-IV CHF;
  * Active liver disease (ALT >2.5 times upper limit of normal);
  * Women who are pregnant;
  * A platelet count of less than 100,000 cells/mm3;
  * Impaired renal function (creatinine ≥2.5 mg/dL) or status post renal transplant;
  * Recipient of heart transplant;
  * Patient with a life expectancy less than 12 months;
  * Known allergies to aspirin, clopidogrel bisulfate (PlavixR) and ticlopidine (TiclidR), heparin, bivalirudin, contrast, or pioglitazone, that cannot be medically managed;
  * Any significant medical condition, which in the investigator's opinion, may interfere with the patient's optimal participation in the study;
  * Currently participating in an investigational drug or another device study;
  * Current use of any thiazolidinedione (Rosiglitazone (Avandia) or Poiglitazone (Actos).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy of rosiglitazone on bare metal stent (BMS) in-stent restenosis measured as late lumen loss in patients with metabolic syndrome.

SECONDARY OUTCOMES:
The secondary parameter for evaluation of efficacy is binary restenosis.
The tertiary objective is to assess the effect of rosiglitazone on major cardiac events and target vessel revascularization).

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States